CLINICAL TRIAL: NCT05089019
Title: An Open-Label, Randomized Study to Evaluate the Bioequivalence of Selpercatinib Formulations
Brief Title: A Study Comparing Two Formulations of Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18177; J2G-MC-JZJZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selpercatinib (Test) (Experimental): 160 mg Selpercatinib (tablet formulation) given orally on days 1 and 15.
  Interventions: Drug: Selpercatinib
- Selpercatinib (Reference) (Active Comparator): 160 mg Selpercatinib (2 X 80 mg capsule formulation) given orally on days 1 and 15.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Administered orally
  Other Names: LY3527723; LOXO-292

SUMMARY:
The main purpose of this study is to compare the amount of selpercatinib that gets into the blood stream and how long it takes the body to get rid of it, when given as different formulations. The information about any adverse effects experienced will be collected and the tolerability of selpercatinib will also be evaluated. The study may last up to 56 days including the 28 days of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and vital signs.
* Participants who have clinical laboratory test results within the normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.

Exclusion Criteria:

* Have a history of allergic reactions to medications or food products
* Have a clinically significant abnormality of blood pressure and/or pulse rate as determined by the investigator
* Clinically significant abnormalities on ECG as determined by the investigator or prolongation of the QTcB or QTcF >450 msec at screening
* Have clinically significant active cardiovascular disease or history of myocardial infarction within 6 months prior to the planned start of selpercatinib
* Have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data. Appendectomy, splenectomy, and cholecystectomy are considered as acceptable
* Use of H2 blockers, proton pump inhibitors, and other drugs that affect selpercatinib exposure within 7 days of screening
* Are intending to use over-the-counter or prescription medication, including dietary supplements, within 14 days prior to dosing and until study discharge (apart from occasional acetaminophen (≤2 g/24 hours), hormonal contraception, or hormone replacement therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - Covance Dallas, Dallas, Texas
  - LabCorp CRU, Inc., Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a washout period of 14 days between doses of selpercatinib.
Groups:
- Sequence 1 - Selpercatinib Reference/Test: Sequence 1: 160 mg selpercatinib (2 x 80 mg capsules) in Period 1, 160 mg selpercatinib (1 x 160 mg tablet) in Period 2.
- Sequence 2 - Selpercatinib Test/Reference: Sequence 2: 160 mg selpercatinib (1 x 160 mg tablet) in Period 1, 160 mg Selpercatinib (2 x 80 mg capsules) in Period 2.
Period: Period 1
Arm/Group | Sequence 1 - Selpercatinib Reference/Test | Sequence 2 - Selpercatinib Test/Reference
Started | 112 | 112
Received at Least One Dose of Study Drug | 112 | 112
Completed | 112 | 111
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period
Arm/Group | Sequence 1 - Selpercatinib Reference/Test | Sequence 2 - Selpercatinib Test/Reference
Started | 112 | 111
Completed | 100 | 104
Not Completed | 12 | 7
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 6 | 3
Period: Period 2
Arm/Group | Sequence 1 - Selpercatinib Reference/Test | Sequence 2 - Selpercatinib Test/Reference
Started | 100 | 104
Received at Least One Dose of Study Drug | 100 | 104
Completed | 95 | 101
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Sequence 1 - Selpercatinib Reference/Test: Sequence 1: 160 mg selpercatinib (2 x 80 mg capsules) Reference/160 mg selpercatinib (1 x 160 mg tablet) Test
- Sequence 2: Selpercatinib Test/Reference: Sequence 2: 160 mg selpercatinib (1 x 160 mg tablet) Test/160 mg selpercatinib (2 x 80 mg capsules) Reference
- Total: Total of all reporting groups
Arm/Group | Sequence 1 - Selpercatinib Reference/Test | Sequence 2: Selpercatinib Test/Reference | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.3) | 42.8 (12.4) | 42.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 59 | 59 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 36 | 71
  Not Hispanic or Latino | 77 | 76 | 153
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 45 | 37 | 82
  White | 59 | 67 | 126
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 112 | 112 | 224

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Selpercatinib
Description: PK: Cmax of Selpercatinib
Time Frame: Day 1 and Day 15: Predose, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 192, 240, and 312 hours (h) postdose;
Population: All participants who received at least 1 dose of Selpercatinib and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 160 mg Selpercatinib (Reference): 160 milligram (mg) Selpercatinib (2 x 80 mg capsules) administered orally on Day 1 or Day 15 according to the randomization schedule.
- 160 mg Selpercatinib (Test): 160 mg Selpercatinib (tablet) administered orally according to the randomization schedule.
Arm/Group | 160 mg Selpercatinib (Reference) | 160 mg Selpercatinib (Test)
Number analyzed (Participants) | 209 | 206
nanograms per milliliter (ng/mL) | 1520 (61) | 1350 (91)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib (Reference) vs 160 mg Selpercatinib (Test); Test type: Equivalence — Equivalence margin 80% to 125%; Mixed Models Analysis; Ratio of Geometric Least Square (LS) Mean; Ratio of Geometric LS Mean = 0.889, 94.12% CI 2-sided [0.810 to 0.976]

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Selpercatinib
Description: PK: AUC[0-∞] of Selpercatinib.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*hr/mL)
Groups:
- 160 mg Selpercatinib (Reference): 160 mg Selpercatinib (2 x 80 mg capsules) administered orally on Day 1 or Day 15 according to the randomization schedule.
Arm/Group | 160 mg Selpercatinib (Reference) | 160 mg Selpercatinib (Test)
Number analyzed (Participants) | 206 | 200
nanograms*hour per milliliter (ng*hr/mL) | 20700 (45) | 19300 (51)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib (Reference) vs 160 mg Selpercatinib (Test); Test type: Equivalence — Equivalence margin 80% to 125%; Mixed Models Analysis; Ratio of Geometric LS Mean = 0.927, 94.12% CI 2-sided [0.882 to 0.975]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Selpercatinib
Description: PK: AUC[0-tlast] of Selpercatinib
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 160 mg Selpercatinib (Testt): 160 mg Selpercatinib (tablet) administered orally according to the randomization schedule.
Arm/Group | 160 mg Selpercatinib (Reference) | 160 mg Selpercatinib (Testt)
Number analyzed (Participants) | 206 | 204
ng*hr/mL | 20200 (47) | 18100 (65)
Statistical Analysis 1: Comparison: 160 mg Selpercatinib (Reference) vs 160 mg Selpercatinib (Testt); Test type: Equivalence — Equivalence margin 80% to 125%; Mixed Models Analysis; Ratio of Geometric LS Mean = 0.891, 94.12% CI 2-sided [0.834 to 0.951]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days
Description: All enrolled participants who received at least one dose of selpercatinib, whether or not they completed all protocol requirements, and have at least one postdose safety assessment.
Groups:
- 160 mg Selpercatinib (2 x 80 mg Reference): 160 mg selpercatinib (2 x 80 mg capsules) will be administered orally on Day 1 and Day 15.
- 160 mg Selpercatinib (1 x 160 mg Test): 160 mg selpercatinib (1 x 160 mg tablet) will be administered orally on Day 1 and Day 15.
Arm/Group | 160 mg Selpercatinib (2 x 80 mg Reference) | 160 mg Selpercatinib (1 x 160 mg Test)
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/212
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/212
Other Adverse Events (participants affected / at risk) | 0/216 | 0/212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT05089019/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT05089019/SAP_001.pdf